CLINICAL TRIAL: NCT03697707
Title: An International, Multicentre, Open-label Study To Evaluate The Efficacy and Safety of Two Different Vaccination Regimens of Immunotherapy With Allogeneic Dendritic Cells, DCP-001, in Patients With Acute Myeloid Leukaemia That Are In Remission With Persistent MRD
Brief Title: Efficacy and Safety of Immunotherapy With Allogeneic Dendritic Cells, DCP-001, in Patients With Acute Myeloid Leukaemia
Acronym: ADVANCE-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mendus (Industry)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCOne-002
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Acute Myeloid Leukemia in Remission
Keywords: AML in CR1 or CRi; DCOne; DCP-001; Minimal Residual Disease
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: First 10 patients will get the lowest dose and next 10 patients will receive the highest dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Low dose (Experimental): patients receiving 4 bi-weekly vaccinations with 25E6 cells/vaccination of DCP-001, and 2 booster vaccinations with 10E6 cells/vaccination
  Interventions: Biological: DCP-001
- Cohort 2: High dose (Experimental): patients receiving 4 bi-weekly vaccinations with 50E6 cells/vaccination of DCP-001, and 2 booster vaccinations with 10E6 cells/vaccination
  Interventions: Biological: DCP-001

INTERVENTIONS:
Biological: DCP-001 — allogeneic dendritic cell vaccine

SUMMARY:
Phase II study to evaluate safety and efficacy of DCP-001 in patients with AML in CR, and with presence of MRD

DETAILED DESCRIPTION:
International, multicentre, open-label proof of concept study exploring two different dose groups of the allogeneic dendritic cell vaccine, DCP-001. Cohort 1 consists of 10 patients that will receive 25E6 DCP-001 cells per vaccination and Cohort 2 consists of 10 patients who will receive 50E6 DCP-001 cells per vaccination. All patients will be given two additional booster vaccinations of 10E6 cells. Each patient will be followed up for 12 months after the 4th vaccination. Safety will be monitored throughout the study. Sera and cell samples (blood and bone marrow) will be collected for assessment of efficacy (MRD evaluation) and immune response monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of AML according to WHO2016 criteria, including cytological, molecular and cytogenetic criteria (except acute pro-myelocytic leukaemia/APL).
2. In CR1 (first complete remission) or CRi (incomplete blood count recovery) documented by bone marrow examination up to one month before vaccination; CR defined as less than 5% blasts in normo-cellular bone marrow, ANC >1*E9/L, platelet count >100*E9/L, no evidence of extra-medullary disease. Patients in CRi (patients with <5% blasts but with incomplete blood count recovery) should have platelets >50 E9/L.
3. MRD as defined by multicolour flow cytometry (MFC) at a value of > 0.1%, or detection of specific molecular abnormalities such as NPM1 mutation.
4. Patients that are in CR1 or CRi. Patients not having undergone consolidation therapy must have been in CR1 for at least 1 month prior to enrolment. Patients treated with hypomethylating agents must have been given at least two cycles and up to a maximum of nine cycles of hypomethylating agents.
5. Expected and willing to undergo all study procedures, including outpatient evaluations for clinical and immunological monitoring.
6. Male or female of ≥ 18 years of age.
7. Women of childbearing potential must be using anti-conceptive therapy or use two (2) barrier contraceptive methods (one by each partner and at least one of the barrier methods must include spermicide (unless spermicide is not approved in the country or region). See section 12.7 for birth control methods deemed acceptable for this study.
8. ECOG (WHO) performance status 0-2.
9. Willing and able to provide written informed consent for participation in the study

Exclusion Criteria:

1. Acute Promyelocytic (APL; M3) type of AML.
2. Patients who have undergone or are scheduled/eligible for allogeneic stem cell transplantation.
3. History of previous allogeneic bone marrow or solid organ transplantation.
4. Uncontrolled or serious infections
5. Ongoing immunosuppressive therapy, other than short use of low dose steroids, i.e. equivalent to an average dose of ≤10mg of prednisone/day.
6. Chemotherapy and antineoplastic hormonal therapy within 28 days prior to the screening visit, with the exception of hypomethylating agents such as azacitidine and decitabine, or midostaurin for FLT3 mutations, or patients treated with IDH12 inhibitors in mIDH1/2.
7. Current or past medical history autoimmune disease.
8. Inadequate liver function (AST and ALT > 3 x ULN, serum bilirubin >3 x ULN).
9. Other active Malignancies within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin or adequately controlled limited basal cell skin cancer.
10. Pregnant or lactating females.
11. Major surgical procedure (including open biopsy) within 28 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment.
12. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (i.e. active) cardiovascular disease.
13. Evidence of any other medical conditions (such as psychiatric illness, physical examination or laboratory findings) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.
14. Known HIV, Hepatitis B and/or Hepatitis C infections.
15. History of hypersensitivity to the investigational medicinal product or to any excipient present in the pharmaceutical form of the investigational medicinal product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
minimal residual disease (MRD) | up to 32 weeks
  Any change in MRD (flow cytometric) as compared to baseline MRD

SECONDARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | up to 56 weeks
  adverse event
Serious Adverse Events (SAEs) | up to 56 weeks
  adverse events
Relapse-free survival | up to 56 weeks
  efficacy
Overall survival | up to 56 weeks
  efficacy
Immune responses | up to 32 weeks
  Any change in immunoreactivity (specific and non-specific) as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: A A van de Loosdrecht, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (10):
- Helsinki University Hospital, Helsinki, Finland
- Germany (4):
  - Universitats Klinikum Bonn, Bonn
  - Marien Hospital, Düsseldorf
  - Universitats Klinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
- Netherlands (3):
  - VUmc, Amsterdam
  - UMCG, Groningen
  - Maastricht University Medical Centre, Maastricht
- Haukeland universitetssjukehus, Bergen, Norway
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] van de Loosdrecht AA, van Wetering S, Santegoets SJAM, Singh SK, Eeltink CM, den Hartog Y, Koppes M, Kaspers J, Ossenkoppele GJ, Kruisbeek AM, de Gruijl TD. A novel allogeneic off-the-shelf dendritic cell vaccine for post-remission treatment of elderly patients with acute myeloid leukemia. Cancer Immunol Immunother. 2018 Oct;67(10):1505-1518. doi: 10.1007/s00262-018-2198-9. Epub 2018 Jul 23. PMID 30039426